CLINICAL TRIAL: NCT01865994
Title: Study to Examine the Correlation of 'Estimated Continuous Cardiac Output' (esCCO) With Transesophageal Echocardiography (TEE) in Pediatric Cardiac Surgery
Brief Title: Correlation of Estimated Continuous Cardiac Output (esCCO) and TEE in Pediatric Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: Nihon Kohden Europe (Unknown)
Responsible Party: Principal Investigator, Christoph Schramm, M.D., Principal Investigator, Heidelberg University
Other Study IDs: S108/2012
Record Dates: First submitted 2013-05-27; First posted 2013-05-31 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Cardiac Diseases Requiring Surgery
Keywords: Cardiac Output; esCCO; TEE; Pediatric cardiac surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pediatric cardiac surgery: Children scheduled for elective cardiac surgery

SUMMARY:
The purpose of this study is to determine the measuring accuracy of the truly non-invasive method estimated continuous cardiac output (esCCO) against the reference method transesophageal echocardiography in pediatric cardiac surgery. esCCO is calculated using the pulse wave transit time, which is defined as the time between the R-wave of the ECG and the 30% increase of the differentiated pulseoximetry waveform.

DETAILED DESCRIPTION:
The objective is to compare two methods of cardiac output measurement in children: the new non-invasive method called esCCO™ (by Nihon Kohden, Tokyo, Japan) and the established more invasive method transesophageal echocardiography (TEE). esCCO™ is a completely non-invasive method that could provide a cardiac output measurement in a large range of pediatric patients because of an extremely low risk benefit balance.

Cardiac output monitoring has been technically challenging in pediatric patients. Available methods for measuring cardiac output in children are either inaccurate or highly invasive or limited to a small number of patients. So far esCCO™ has not been tested in the pediatric population but showed promising results when it was tested against the pulmonary artery catheter in adult patients undergoing heart surgery in previous Japanese studies.

Thus the validity of esCCO™ is now tested in pediatric patients scheduled for elective cardiac surgery. Transesophageal echocardiography has been chosen as reference method because it is performed routinely during pediatric cardiac surgery.

The algorithm for esCCO™ -measurement is integrated in an approved patient monitor that replaces the standard patient monitor during the measurement-period.

In the study protocol, events like esCCO™ -calibration time, catheter positioning time, ventilation settings, volume in- and output and drug administration, patients's data and diagnoses are logged. Vital parameters from the patient monitor including the esCCO™-cardiac output values are recorded every second in real time on a study laptop mounted on the same rack as the patient monitor but electrically separated from the other devices.

EsCCO™ measurements shall be compared to TEE cardiac output measurements at three given times: (1) before surgical intervention, (2) shortly after cardiopulmonary bypass and (3) after closure of the thorax.

A total of 50 patients shall be investigated in the study during a planned study time of approximately 6 months. The ethics committee of the University of Heidelberg gave their consent to the study (S-108/2012). For statistical analysis, a Bland-Altman-test for measurements with multiple values per patient, correlation graphics and a regression equation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* children <=18 years
* elective cardiac surgery
* Sinus rhythm

Exclusion Criteria:

* no written consent
* continuous severe cardiac arrhythmias
* cardiac Pacemaker
* intraaortal balloon pump
* contraindications for TEE
* persistent ductus arteriosus botalli

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients (0-18 yrs) scheduled for elective cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2012-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | Intraoperative
  EsCCO™ measurements shall be compared to TEE cardiac output measurements at three given times: (1) before surgical intervention, (2) shortly after cardiopulmonary bypass and (3) after closure of the thorax

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Heidelberg, Germany